CLINICAL TRIAL: NCT06250894
Title: A Clinical Study of the Efficacy and Safety of Sintilimab in Combination With Chemotherapy (S-1/Oxaliplatin, SOX) and Radiotherapy for the Neoadjuvant Treatment of Locally Advanced Esophagogastric Junction Adenocarcinoma
Brief Title: Neoadjuvant Sintilimab Plus Chemoradiotherapy for Locally Advanced Adenocarcinoma of Esophagogastric Junction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018S00686
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: PD-1; Neoadjuvant Chemoradiotherapy; Gastroesophageal Junction Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant immunotherapy-chemoradiotherapy (Experimental): This is a one arm study, enrolled locally advanced EGJ patients will receive Sintilimab (PD-1 inhibitor) and combined with preoperative chemoradiotherapy and operation.
  generic name：PD-1; dosage form：Injection; dosage：200mg (20ml)； frequency：every 3 weeks； duration：3 times before operation and 3-5 times after operation
  Interventions: Drug: PD-1inhibitor

INTERVENTIONS:
Drug: PD-1inhibitor — Patients receive 3 cycles of preoperative chemotherapy with Sintilimab（PD-1 inbibitor） and SOX (every 3 weeks), followed by radiotherapy (total dose of 36-40Gy in 18-22 fractions) during cycle 1 of the combination. Radical surgery for gastric cancer will be performed within 4-6 weeks after completion of neoadjuvant treatment, followed by 3-5 cycles of postoperative adjuvant chemotherapy with the SOX regimen.

SUMMARY:
The purpose of this study is to access the safety and efficacy of neoadjuvant Immunotherapy (Sintilimab, PD-1 inhibitor) combined with chemotherapy (S-1+Oxaliplatin) and radiotherapy for locally advanced esophagogastric junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70, male and female.
* Histologically confirmed locally advanced esophagogastric junction Adenocarcinoma cT3-4aNxM0 (AJCC v8), Siewert typed as type II-III.
* No previous anti-tumor treatment.
* ECOG score was 0-1.
* Expected survival of ≥ 6 months
* Adequate organ reserve function.

Exclusion Criteria:

* Malignant disease other than gastric cancer (excluding radically treated basal cell carcinoma of the skin, squamous epithelial carcinoma of the skin, and/or radically resected carcinoma in situ) diagnosed within 5 years.
* Known Her-2 positive( IHC 3+ or FISH positve).
* Patients have received immunotherapy, such as PD-1 antibody, PD-L1 antibody and CTLA4 antibody
* Severe allergic reaction to monoclonal antibody.
* Receiving systemic glucocorticoid therapy within 7 days prior to the first dose of the study
* Known endoscopic signs of active bleeding from the lesion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response | 10 days after operation
  No malignant tumor cells were detected in the removed specimens including primary tumor and lymph nodes

SECONDARY OUTCOMES:
Objective response rate (ORR) | 6 months after the recruitment of the last subject.
  The Objective response rate (ORR) is defined as the proportion of patients with a complete response (CR) or a partial response (PR) to preoperative therapy. The ORR will be evaluated using the RESIST1.1 protocol.
Disease-Free-Survival (DFS) | Through study completion, an average of 1 year
  The time between the beginning of treatment and the observation of disease progression or death from any cause.
Number of participants with AEs (Adverse Events) | Through study completion, an average of 1 year
  The AEs during the trial, including radiation mucositis, bone marrow suppression, AEs related to immunotherapy and so on. The AEs will be evaluated using the CTCAE 5.0 protocol.
Major pathologic response (MPR) | 10 days after operation
  defined as residual tumors less than 10% after neoadjuvant immunotherapy and(or) chemotherapy
Overall survival (OS) | Through study completion, an average of 1 year
  OS was the time from enrolment to death from any cause. OS was censored on the last date known to be alive for patients without documentation of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Min Jin, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No